CLINICAL TRIAL: NCT01383070
Title: Effectiveness of Cell Phone Counseling to Improve Breast Feeding Indicators
Brief Title: Evaluation of Effectiveness of Cell Phone Technology as Community Based Intervention to Improve Exclusive Breast Feeding
Acronym: BFC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lata Medical Research Foundation, Nagpur (Other)
Responsible Party: Dr. Archana Patel, Principal Investigator, CEO and Vice President, Lata Medical Resarch Foundation, Nagpur
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01_BFC
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Malnutrition in Pregnancy; Other Disorders of Breast and Lactation Associated With Childbirth
Keywords: Timely initiation of breast feeding; Exclusive breast feeding; Timely introduction of complimentary feeding; Breast Feeding, Exclusive; Childbirth and the Puerperium
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactational Conseling (No Intervention): The existing staff of the hospitals will be provided training in IYCF by BPNI. They will be encouraged to set up their own systems to continue counseling during the ante natal period, at delivery and during the immunization visits. The participants will be asked to come for the same schedule of visits as in the intervention group where their data will be collected.
  Interventions: Behavioral: Lactational Counseling by Cell phone
- Lactation Counseling by Cell Phone (Experimental): The approach to promoting TIBF, EBF and TICF will be through cell phone counseling in addition to counseling in the hospitals during scheduled ante natal visits. Mother in the intervention group (beneficiaries) would be provided handsets and included in a subsidized calling plan.
  Interventions: Behavioral: Lactational Counseling by Cell phone

INTERVENTIONS:
Behavioral: Lactational Counseling by Cell phone — The approach to promoting TIBF, EBF and TICF will be through cell phone counseling in addition to counseling in the hospitals during scheduled ante natal visits. Mother in the intervention group (beneficiaries) would be provided handsets and included in a subsidized calling plan.
  Other Names: Cell Phone Counseling; Lactational Counseling

SUMMARY:
Primary hypotheses

In a hospital-based CRCT, cell phone lactational counseling starting in the third trimester of pregnancy to 24 weeks after delivery will improve the prevalence of EBF by 7.5 % (7.5% increase in EBF by retraining in BFHI alone in both groups from baseline and a additional 7.5% improvement in intervention group as compared to the control) compared with women with from hospitals with only retraining BFHI.

Secondary hypotheses As compared to women from hospitals receiving only retraining in BFHI, those with additional cell phone lactational counseling will experience the following

* Increase in the percentage of EBF(breast milk and no other foods or milk based liquids) at 24 weeks after delivery,
* Increase in the mean duration of any breastfeeding,
* Increase in the percentage with TIBF,
* Reduction in use of pre lacteal feeds
* Reduction in percentage of infants being bottle fed(any liquid or semi-solid food from a bottle with nipple/teat) any time before or at 24 weeks
* Increase in the percentage of infants at 26 weeks after delivery who receive TICF,
* Increase in growth velocity (weight, length and head circumference)
* Reduction in the number hospitalizations or mortality in the mother-infant dyad till 26 weeks after delivery
* Increase in adherence to visit schedules
* Greater ratio of effectiveness as compared to costs incurred for cell phone counseling.

DETAILED DESCRIPTION:
Pre Intervention phase- Baseline data regarding breastfeeding parameters will be collected from the participating hospitals in the pre-intervention phase of 3 months. Training in BFHI principles will be conducted at all the participating hospitals by BPNI.

Intervention plan- The interventions will be delivered to the women in the intervention cluster starting in pregnancy and until their child is 26 weeks to finally evaluate the TICF.

a. Description of intervention The approach to promoting TIBF, EBF and TICF will be through cell phone counseling in addition to counseling in the hospitals during scheduled ante natal visits. Mother in the intervention group (beneficiaries) would be provided handsets and included in a subsidized calling plan.

i) Selection and training of cell phone LCs Motivated women with personal breastfeeding experience with at least a diploma in nursing will be recruited and trained in person-to-person and tele-counseling. Counseling skills will be taught mainly by demonstrations and role play and will include: how to communicate, listen to mothers, learn about their difficulties, build mother's confidence, give support and providing relevant information and practical help when required. BPNI will conduct the 51 hour "An integrated course on Breastfeeding, Complementary feeding and Infant Feeding & HIV - Counseling" with clinical practice in the ante natal and post natal counseling with pregnant women and mothers in the hospitals.

ii) Counseling schedules: There will be personal counseling(based on the BPNI training) during scheduled hospital visits: 2 in the antenatal period, 1 at the time of delivery and then during immunization visits at 6, 10 and 14 weeks, at 24 weeks and at the end of 26 weeks post natal. The participants will be free to make additional visits if they need medical attention.

Antenatal visits: During the two antenatal contacts the counselors will prepare the mothers, and other members of the family who will support her at delivery how to initiate breastfeeding within one hour of delivery. They will discourage prelacteal feeds and other fluids and foods after lactation has been initiated. They will encourage the mothers to eat more of their usual foods to support enhanced lactation, and to appropriately rest during the third trimester. These meetings will also cover problems with breastfeeding that the mother might encounter and how best to deal with them.

At delivery: The messages to promote TIBF and EBF will be reinforced. Post Natal Visits (6, 10, and 14, 24 and 26 weeks): The mothers will visit the hospital for the scheduled immunization visits where they will be inquired if they have any difficulties in feeding the infant. They will be referred to the LCs if they have difficulties. Data will be collected from her regarding the IYCF practices, illnesses of mother and child necessitating hospitalization, maternal satisfaction regarding IYCF counseling, cost data in standardized case report forms. She will be encouraged to talk to the LCs on cell phone for any issues about IYCF between 2 visits.

iii) Tele Counseling: It is anticipated that each counselor will be able to support 10 calls a day. The duration of each call could vary according to the problem from 10 to 30 minutes. LCs will be taught how to respond to the phone calls by role playing and practice sessions with a number of problems that a mother can encounter. The calls will be recorded on the mobile and the voice data will be transferred from the handset to the computer. The confidentiality and anonymity of the caller will be maintained. Each LC and cell phone user will be trained by the Vodafone Essar trainers (mobile carrier which has partnered with us in this project) on how to use and handle the handsets, for outgoing calls, incoming calls, short messages and how to charge the phones. The counselor's numbers will be on speed dial and the beneficiaries and the LCs will be within one caller group. All incoming messages and calls would be free of charge to the beneficiary. Recharge option will be made available. All beneficiaries will receive short messages daily in their vernacular language, and scheduled weekly calls from the LCs. They will also be sent messages to adhere to their schedules. Additionally they can also call the LCs when they have difficulties in feeding their infant. The calls will begin from the time they enroll till their last scheduled visit. Ringtones to encourage breast feeding will also be provided. They would be encouraged to call between 9 am to 6 pm unless it is an emergency.

ELIGIBILITY:
Inclusion Criteria:

* Mother's registered at the antenatal clinic at 32-36 weeks gestation and planning to deliver in the same hospital and willing to follow up at the same hospital till 26 weeks infant age.
* Absence of illness that will interfere with EBF - severe anemia (Hb < 6); eclampsia, pre-eclampsia, mother needing medicine for which breastfeeding is contraindicated, HIV positivity
* living in catchment area of 20 km from hospital.

Exclusion Criteria:

* Those who do not fulfill inclusion criteria

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1036 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Changes in the percentage of women exclusively breastfeeding (breast milk and no other foods or milk based liquids) their infants at 24 weeks. | 26th week after delivery
  Measurement: Maternal recall of infant feeding practices over last 24 hrs will be elicited with a structured questionnaire at 24 weeks infant age. The infant receiving only breastmilk and no supplemental liquids or solid foods other than vitamins, minerals supplements or medicines in last 24 hrs will be considered to be EBF.

SECONDARY OUTCOMES:
Growth through 6 months of age - weight, length and head circumference gains between birth and each immunization visit (at 6, 10 and 14 weeks), at 24 weeks and at 26 weeks for growth velocity. | 26th week after Delivery
  Unclothed weight will be measured using digital electric scales to the nearest 1g. Supine length will be measured using a infantometer to the nearest 0.5 cm. Occipito-frontal head circumference will be measured using a non-stretchable tape; mean of three measurements will be taken. Training will be provided for all measurement techniques and performance will be assessed at regular intervals during the study. Scales and infantometers will be calibrated regularly against standards at all sites.

CONTACTS AND LOCATIONS:
Overall Officials: Archana B Patel, MD,DNB,PhD, Principal Investigator — CEO and Vice President, LMRF And Professor & Head Pediatrics, Indira Gandhi Govt. Medical College, Nagpur
Locations (1):
- Lata Medical Research Foundation, Nagpur, Nagpur, India